CLINICAL TRIAL: NCT01324960
Title: A Phase I and Phase II Study of the Efficacy and Safety of Maintenance Treatment With Azacitidine With or Without Ceplene/Interleukin-2 in Patients With Higher Risk Myelodysplastic Syndromes Who Achieved Hematological Response to Azacitidine
Brief Title: Azacitidine With or Without Ceplene/Interleukin-2 in Patients With Higher Risk Myelodysplastic Syndromes
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Groupe Francophone des Myelodysplasies (Other)
Collaborators: EpiCept Corporation (Industry)
Responsible Party: Céline Berthon, MD, Groupe Francophone des Myelodysplasies
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GFM-Aza-ceplene
Record Dates: First submitted 2011-03-07; First posted 2011-03-29 (Estimated); Last update posted 2014-03-20 (Estimated); Status verified 2011-03

CONDITIONS: Myelodysplastic Syndromes
Keywords: IPSS; High risk; Azacitidine; Ceplene
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Histamine; Interleukin-2; Azacitidine; lactitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ceplene® / IL2 + Azacitidine (Experimental): Azacitidine 75 mg/m2 subcutaneously daily for 7 days every 4 weeks. Ceplene® / IL2: Patients will receive Ceplene (EpiCept Corporation, Tarrytown, NY) at 0.5 mg subcutaneous twice daily and human recombinant IL-2 (aldesleukin; Novartis) 16 400 U/kg subcutaneous twice daily during 15 days for up to 10 cycles, on days 8 to 21 of AZA cycles.
  Interventions: Drug: Ceplene®, IL-2, Azacitidine
- Azacitidine (Active Comparator): Azacitidine 75 mg/m2 subcutaneously daily for 7 days every 4 weeks
  Interventions: Drug: Azacitidine

INTERVENTIONS:
Drug: Ceplene®, IL-2, Azacitidine — Azacitidine: 75 mg/m2 subcutaneously daily for 7 days every 4 weeks. Ceplene® / IL2: Patients will receive Ceplene at 0.5 mg subcutaneous twice daily and human recombinant IL-2 at 16 400 U/kg subcutaneous twice daily during 15 days for up to 10 cycles, on days 8 to 21 of AZA cycles.
  Other Names: Human recombinant IL-2 = Aldesleukin® (Novartis); Azacitidine = Vidaza® (Celgene)
  Arms: Ceplene® / IL2 + Azacitidine
Drug: Azacitidine — Azacitidine 75 mg/m2 subcutaneously daily for 7 days every 4 weeks
  Other Names: Azacitidine = Vidaza® (Celgene)
  Arms: Azacitidine

SUMMARY:
A phase I study of azacitidine with Ceplene/interleukin-2 will first evaluate the safety and tolerability of this regimen in patients with higher risk myelodysplastic syndromes (MDS) who achieved a hematological response after 6 cycles of azacitidine. After approval by an independent Data Safety Monitoring Board (DSMB), the phase I study will be followed by an open label randomized phase II study designed to characterize the efficacy, safety, and tolerability of the addition of Ceplene/interleukin-2 to azacytidine in patients with higher risk myelodysplastic syndrome (MDS) who achieved a hematological response after 6 cycles of azacitidine.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Must understand and voluntarily sign an informed consent form
* Must be able to adhere to the study visit schedule and other protocol requirements
* Documented diagnosis of MDS according to WHO classification, that meets IPSS criteria for intermediate-2 or high-risk disease
* Must have achieved a response (CR, PR, mCR or HI according to IWG 2006 criteria) after 6 cycles of Azacitidine.
* Patients must have ECOG performance status (PS) of 0 - 2.
* Women of child-bearing potential (i.e., women who are pre-menopausal or not surgically sterile) must have a negative serum or urine pregnancy test within 2 weeks prior to beginning treatment on this study. Nursing patients are excluded.
* Creatinine clearance >50 ml/min
* Serum aspartate aminotransferase (AST)/serum glutamic-oxaloacetic transaminase (SGOT) or alanine transaminase (ALT)/serum glutamate pyruvate transaminase (SGPT) < 3.0 x upper limit of normal (ULN)
* Serum total bilirubin < 1.5 mg/dL. (except for unconjugated hyperbilirubinemia due to Gilbert's disease or secondary to MDS).

Exclusion Criteria:

* Known positive status for human immunodeficiency virus (HIV) or hepatitis B or C
* Uncontrolled intercurrent illness including, but not limited to uncontrolled infection, symptomatic congestive heart failure, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients receiving any other standard or investigational cytotoxic treatment for their hematologic malignancy
* Any medical condition which in the opinion of the investigator places the patient at an unacceptably high risk for toxicities
* Prior history of malignancy other than MDS (except basal cell or squamous cell carcinoma or carcinoma in situ of the cervix or breast) unless the subject has been free of disease for ≥ 3 years
* Class III or IV cardiac disease, hypotension or severe hypertension, vasomotor instability, serious or uncontrolled cardiac dysrhythmias (including ventricular arrhythmias) at any time, acute myocardial infarction within the past 12 months, active uncontrolled angina pectoris or symptomatic arteriosclerotic blood vessel disease
* History of seizures, central nervous disorders, stroke within the last 12 months, or psychiatric disability thought to be clinically significant in the opinion of the investigator
* Prior history of autoimmune disease (including but not limited to systemic lupus, inflammatory bowel disease, and psoriasis)
* Patients with active peptic or esophageal ulcer disease or with past peptic ulcer or esophageal disease with a history of bleeding
* Patients continuing systemic treatment with clonidine, steroids, and/or H2 receptor blocking agents Patients with a history of hypersensitivity to histamine or histamine products, severe allergies to food or contrast media requiring treatment within the last five years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-03; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Time to progression according to IWG2006 criteria | Every 4 cycles (during average 2 years)
  Progression will be assessed by monitoring the bone marrow, blood and hematologic supportive care according IWG 2006 criteria .

SECONDARY OUTCOMES:
Types and numbers of adverse events occuring in all treated patients | Every cycle, during the follow-up on average during 2 years
  The safety profile will be determine by assessements of clinical symptoms, physical examinations, vital signs and clinical laboratory tests. The types and numbers of adverse events occuring in all treated patients will be tabulated.
Improvement of the quality and the duration of responses compared to maintenance with AZA alone | While patient is on study, during follow up on average during 2 years
  The response will be assessed every 4 cycles according IWG 2006 criteria and it will be evaluated if there is an improvement of the level of response and the response duration

CONTACTS AND LOCATIONS:
Overall Officials: Céline BERTHON, MD, Principal Investigator — Groupe Francophone des Myelodisplasies; Bruno QUESNEL, MD, PhD, Principal Investigator — Groupe Francophone des Myelodisplasies; Pierre Fenaux, MD, Principal Investigator — Groupe francophone des Myelodisplasies
Locations (28):
- France (28):
  - CHU d'Amiens, Amiens
  - CHU Angers, Angers
  - CH d'Avignon, Avignon
  - Hôpital de la Côte Basque, Bayonne
  - Hopital Avicenne, Bobigny
  - CHU de Caen, Caen
  - CHU de, Clermont-Ferrand
  - Centre Hospitalier Sud-Francilien, Corbeil-Essonnes
  - CHU Grenoble, Grenoble
  - Hôpital Versailles, Le Chesnay
  - Hôpital Saint Vincent, Lille
  - CHRU Hurriez, Lille
  - CHRU Limoges, Limoges
  - Hôpital Edouard Heriot, dpt Hématologie Clinique, Lyon
  - Hôpital Paoli-Calmettes, Marseille
  - Hematology Dpt, Hopital de l'Hotel Dieu, Nantes
  - CHU Archet, Nice
  - Hopital Saint Louis, Paris
  - Hôpital Saint Antoine, Paris
  - Centre Hospitalier Joffre, Perpignan
  - Hôpital Jean-Bernard, Poitiers
  - CHRU de Reims, Reims
  - Centre Henri Bequerel, Rouen
  - Centre Hospitalier Universitaire de STRASBOURG, Strasbourg
  - Hopital Purpan Service d'Hématologie Clinique, Toulouse
  - Hopital Bretonneau, Tours
  - CHU de Bicêtre, Le Kremlin-Bicêtre, Île-de-France Region
  - CHU Cochin, Paris, Île-de-France Region